CLINICAL TRIAL: NCT05604768
Title: Study on the Initiation and Immunological Mechanism of Parturition
Brief Title: Study on Initiation and Immunological Mechanism of Childbirth
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Wei Yi, Director, Head of Obstetrics and Gynecology, Beijing Ditan Hospital
Other Study IDs: KY2022-03
Record Dates: First submitted 2022-10-14; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Pregnancy
Keywords: Parturition; Immunity; Myelogenous suppressor cells; Fetal free DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal parturient group: 20 normal parturients who had undergone antenatal examination and delivery in Beijing Ditan Hospital were fully informed of the risks and volunteered to join the study and signed the informed consent form.
- Pregnant women with threatened premature delivery group: 20 pregnant women with threatened preterm labor who had undergone antenatal examination and delivery in Beijing Ditan Hospital were fully informed of the risks and volunteered to join the study and signed the informed consent form.

SUMMARY:
This study is a prospective observational study. The participants including 40 pregnant women who have been filed and delivered in our hospital will enrolled, collect venous blood will be collected at different stages of pregnancy, delivery, postpartum to detect the concentration of fetal free DNA, the frequency of associated immune cells, and the expression of functional molecules, so as to explore the immunological mechanism of delivery initiation.

DETAILED DESCRIPTION:
This study is a prospective observational study. The participants including 40 pregnant women (20 normal parturients and 20 pregnant women with threatened preterm delivery) who have been filed and delivered in our hospital will enrolled, collect venous blood will be collected before 12 weeks of pregnancy, at 24 weeks of pregnancy, at 36 weeks of pregnancy, during parturition, and at 42 days after delivery to conduct the following research: 1) Studying the frequency of peripheral blood MDSCs, pDC and NK cells and the expression of functional molecules at different stages of pregnancy (12,24,36 weeks of pregnancy), before delivery and 42 days after delivery through the expression of relevant functional molecules. 2) Detecting the levels of cytokines and chemokines in peripheral blood at different stages of pregnancy (12,24,36 weeks of pregnancy), before delivery and 42 days after delivery, including: IL-1 β, IL-6, IL-10, IL-18, TGF- β and TNF- α, GM-CSF , IL-23, IL-17, IL-13, IL-4, IL-2, IFN-, IFN-, IL-8, GRO α, GCSF, GMCSM, CCL2, CCL5, CCL26,CXCL8, CXCL12，PGE2, M-CSF, COX2, CCL3, CCL4, CXCL1, IDO, Arg-1, ROS and NO. 3) Detection of cffDNA concentration in peripheral blood at different stages of pregnancy (12,24,36 weeks of pregnancy), before delivery and 42 days after delivery. 4) Detection of frequency of MDSCs, pDC and NK cells and expression of functional molecules in placenta. 5) Frequency of peripheral blood MDSCs, pDC and NK cells, expression of functional molecules, cytokine level and cffDNA concentration in pregnant women with threatened preterm labor. 6) Collecting and studying the demographic data of pregnant women at different stages of pregnancy (12,24,36 weeks of pregnancy), before delivery and 42 days after delivery, adverse events of mothers and infants in the perinatal period, and auxiliary examination data (blood routine test, liver and kidney function, TSH, infection index of Aimei B and C, TSH, blood glucose, blood coagulation function, estrogen and progesterone levels, ultrasound, electrocardiogram, etc).

ELIGIBILITY:
Inclusion Criteria:

* 20 normal parturients and 20 pregnant women with threatened preterm labor who had undergone antenatal examination and delivery in Beijing Ditan Hospital were fully informed of the risks and volunteered to join the study and signed the informed consent form.

Exclusion Criteria:

* 1. Combined with HCV, HIV, syphilis or other infectious diseases.
* 2. Chronic diseases such as diabetes, hypertension, thyroid disease and autoimmune disease.
* 3. Both husband and wife or their families have delivered congenital abnormal fetus in the past.
* 4. Either spouse is unwilling to participate in this study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 20 normal parturients and 20 pregnant women with threatened preterm labor who had undergone antenatal examination and delivery in Beijing Ditan Hospital were fully informed of the risks and volunteered to join the study and signed the informed consent form.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-03-28 (Estimated); Study Completion 2025-03-28 (Estimated)

PRIMARY OUTCOMES:
The change of the frequency of myeloid-derived suppressor cells (MDSCs) in normal pregnancy and delivery | at 12 weeks of pregnancy, at 24 weeks of pregnancy, at 36 weeks of pregnancy, at parturition, and at 42 days after delivery
  The frequency of MDSCs in maternal blood and placenta during normal pregnancy and delivery.
The change of functional molecules expression of myeloid-derived suppressor cells (MDSCs) in normal pregnancy and delivery | at 12 weeks of pregnancy, at 24 weeks of pregnancy, at 36 weeks of pregnancy, at parturition, and at 42 days after delivery
  The expression of functional molecules of MDSCs in maternal blood and placenta during normal pregnancy and delivery.
The change of the frequency of plasmacytoid dendritic cells (pDC) in normal pregnancy and delivery | at 12 weeks of pregnancy, at 24 weeks of pregnancy, at 36 weeks of pregnancy, at parturition, and at 42 days after delivery
  The frequency of pDC in maternal blood and placenta during normal pregnancy and delivery.
The change of the functional molecules expression of plasmacytoid dendritic cells (pDC) in normal pregnancy and delivery | at 12 weeks of pregnancy, at 24 weeks of pregnancy, at 36 weeks of pregnancy, at parturition, and at 42 days after delivery
  The expression of functional molecules of pDC in maternal blood and placenta during normal pregnancy and delivery.
The change of the frequency of Nature Killer (NK) cells in normal pregnancy and delivery | at 12 weeks of pregnancy, at 24 weeks of pregnancy, at 36 weeks of pregnancy, at parturition, and at 42 days after delivery
  The frequency of NK cells in maternal blood and placenta during normal pregnancy and delivery.
The change of the functional molecules expression of Nature Killer (NK) cells in normal pregnancy and delivery | at 12 weeks of pregnancy, at 24 weeks of pregnancy, at 36 weeks of pregnancy, at parturition, and at 42 days after delivery
  The expression of functional molecules of NK cells in maternal blood and placenta during normal pregnancy and delivery.
The change of the content of cffDNA in normal pregnancy and delivery | at 12 weeks of pregnancy, at 24 weeks of pregnancy, at 36 weeks of pregnancy, at parturition, and at 42 days after delivery
  The content of cffDNA in maternal blood and placenta during normal pregnancy and delivery.

SECONDARY OUTCOMES:
The change of the frequency of myeloid-derived suppressor cells (MDSCs) in Pregnant women with threatened premature delivery | at 12 weeks of pregnancy, at 24 weeks of pregnancy, at 36 weeks of pregnancy, at parturition, and at 42 days after delivery
  The frequency of MDSCs in maternal blood and placenta in Pregnant women with threatened premature delivery.
The change of functional molecules expression of myeloid-derived suppressor cells (MDSCs) in Pregnant women with threatened premature delivery | at 12 weeks of pregnancy, at 24 weeks of pregnancy, at 36 weeks of pregnancy, at parturition, and at 42 days after delivery
  The expression of functional molecules of MDSCs in maternal blood and placenta in Pregnant women with threatened premature delivery.
The change of the frequency of plasmacytoid dendritic cells (pDC) in Pregnant women with threatened premature delivery | at 12 weeks of pregnancy, at 24 weeks of pregnancy, at 36 weeks of pregnancy, at parturition, and at 42 days after delivery
  The frequency of pDC in maternal blood and placenta in Pregnant women with threatened premature delivery.
The change of functional molecules expression of plasmacytoid dendritic cells (pDC) in Pregnant women with threatened premature delivery | at 12 weeks of pregnancy, at 24 weeks of pregnancy, at 36 weeks of pregnancy, at parturition, and at 42 days after delivery
  The expression of functional molecules of pDC in maternal blood and placenta in Pregnant women with threatened premature delivery.
The change of frequency of Nature Killer (NK) cells in Pregnant women with threatened premature delivery | at 12 weeks of pregnancy, at 24 weeks of pregnancy, at 36 weeks of pregnancy, at parturition, and at 42 days after delivery
  The frequency of NK cells in maternal blood and placenta in Pregnant women with threatened premature delivery.
The change of functional molecules expression of Nature Killer (NK) cells in Pregnant women with threatened premature delivery | at 12 weeks of pregnancy, at 24 weeks of pregnancy, at 36 weeks of pregnancy, at parturition, and at 42 days after delivery
  The expression of functional molecules of NK cells in maternal blood and placenta in Pregnant women with threatened premature delivery.
The change of the content of cffDNA in Pregnant women with threatened premature delivery | at 12 weeks of pregnancy, at 24 weeks of pregnancy, at 36 weeks of pregnancy, at parturition, and at 42 days after delivery
  The content of cffDNA in maternal blood and placenta in Pregnant women with threatened premature delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Yi, Doctor, Study Director — Beijing Ditan Hospital
Locations (1):
- Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality, China